CLINICAL TRIAL: NCT04810143
Title: Development of an Assay for Tacrolimus Blood Trough Measurement in Pediatric Heart Transplant Patients Using Volumetric Absorptive Microsampling (VAMS) and Stable-Labeled Isotope Dilution Tandem Mass Spectrometry.
Brief Title: Tacrolimus Microsampling
Acronym: VAMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2019-0943
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Validate Volumetric Absorptive Microsampling (VAMS) Assay

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Aim 1 (Experimental): All patients presenting for routine post-transplant care including, but not limited to: cardiac catheterization, cardiac biopsy, inpatient admission, or outpatient visits. A convenience sample of 25 inpatient samples will be collected for Aim 1. Although the assay developed by the MSCF will be validated for accuracy, the purpose of Aim 1 is to test "real world" application of the Mitra Microsampler tubes against the gold standard of blood collected by venipuncture in a controlled setting. To accomplish this, consecutive inpatient heart transplant patients will be enrolled. That sample will be collected at the same time (+/- 15 minutes) as a clinically-indicated, appropriately-timed venipuncture for measurement of a tacrolimus trough and prior to the subject taking tacrolimus so as to represent a trough.
  Interventions: Device: Mitra Microsampler
- Aim 2 (Experimental): Outpatient. A convenience sample of 25 outpatients collecting 1-2 samples will be collected for Aim 2. For those who agree to participate, the parent/patient will be taught by a member of the team on how to use the Microsampler to collect blood from a finger stick. They will be provided with a kit for collection of up to 2 samples and will also be provided with appropriate shipping materials to return samples to CCHMC. Participants will then be instructed to collect a sample in the Mitra Microsampler via fingerstick. In addition to the process of collecting the sample in Aim 2, appropriately-aged participants and/or families will be asked to fill out a brief survey regarding sample collection. This will include questions about the ease or difficulty of performing the steps and tolerability of the procedure relative to past experiences with values obtained by venipuncture.
  Interventions: Device: Mitra Microsampler

INTERVENTIONS:
Device: Mitra Microsampler — an FDA Class I medical device for direct specimen collection of blood or other biological fluids

SUMMARY:
This is a feasibility study at a single site, Cincinnati Children's Hospital Medical Center. Patients who have undergone heart transplantation who meet eligibility requirements will be approached to participate in the study. The purpose of this study is to establish a reliable, home-based method for collecting samples as well as a standardized method for use of small-volume samples on both inpatients and outpatients.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric, adolescent, or young adult patients ≥1 and ≤21 years of age

   1. Aim 1: All patients presenting for routine post-transplant care including, but not limited to: cardiac catheterization, cardiac biopsy, inpatient admission, or outpatient visits
   2. Aim 2: outpatient
2. Currently taking tacrolimus

Exclusion Criteria:

1. Non-English-speaking patients
2. Unable to access overnight delivery services (Aim 2 only)

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Accuracy of +/-10% | 18-24 months from start of enrollment
  A VAMS-based tacrolimus trough values will be accurate +/-10% when compared with standard whole blood values achieved via venipuncture.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Ryan, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided